CLINICAL TRIAL: NCT06041295
Title: Interprofessional Collaborative Practice Between Respiratory Therapists and Nurses- Quality Improvement Project of the Correct Rate of Nurse Guiding Incentive Spirometry After Cardiac Surgery
Brief Title: Quality Improvement Project of Nurse Guiding Incentive Spirometry After Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202308062RINB
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Lung Expansion Therapy; Post-cardiac Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the cardiovascular surgery ICU nurse staff (Experimental): on-the-job training of lung expansion therapy
  Interventions: Behavioral: on-the-job training of lung expansion therapy

INTERVENTIONS:
Behavioral: on-the-job training of lung expansion therapy — on-the-job training of lung expansion therapy

SUMMARY:
Studies have shown that patients undergoing general anesthesia surgery are prone to pulmonary complications after surgery; about 30-72% of cardiac surgery patients have postoperative chest X-rays that reveal lung collapse, leading to gas exchange disorders and hypoxemia. Postoperative lung expansion therapy can increase ventilation-perfusion balance, increase lung volume, promote respiratory mucosal sputum production and reduce postoperative pain, and has been proven to improve postoperative pulmonary-related complications.

Inducement spirometry is currently one of the mainstream methods of performing lung expansion treatment. It uses visual feedback to allow the patient to perform slow, deep breathing with sufficient airflow or volume to achieve the lung expansion effect; it is also used after cardiac surgery in our hospital. The main way for patients to perform lung expansion therapy; compared with only performing respiratory exercises after surgery, induced spirometry can reduce the incidence of lung collapse and respiratory distress in postoperative patients, and can also shorten the ICU stay and total hospitalization stay.

Most cardiac surgery patients in our hospital are given health education on lung expansion therapy by nursing staff before and after surgery. This unit does not have specialized courses on lung expansion therapy, which may lead to differences in explanations between different nursing staff; some patients' lack of knowledge and understanding of lung expansion treatment resulted in the treatment effect not being as good as expected, which motivated the author to formulate a project for improvement. We hope to analyze, review and improve the current situation to improve the effectiveness of lung expansion treatment for patients.

Based on the current situation analysis and relevant literature, a project to improve nursing guidance for lung expansion therapy was implemented.

DETAILED DESCRIPTION:
The following options were selected as solutions:

1. Develop Inducement Spirometry Care Standards
2. Organize in-service education courses on pulmonary dilatation therapy for nursing staff
3. Make a health education leaflet on incentive spirometer and place it in the ward for patients to read.
4. Provide demonstration materials for nursing staff to experience the treatment process

The main purposes are:

1. Improve nursing staff's awareness of lung expansion therapy
2. Improve the accuracy of nursing staff in performing lung expansion therapy and health education
3. Improve the accuracy of patients' lung expansion therapy
4. Reduce the incidence of pulmonary complications in patients after cardiac surgery

ELIGIBILITY:
Nurses:

Inclusion Criteria:

* Nurse staff in cardiovascular surgery ICU of National Taiwan University Hospital

Exclusion Criteria:

* None

Patients:

Inclusion Criteria:

* 18 years of age and above
* Perform cardiovascular surgeries at National Taiwan University Hospital
* After surgery, the endotracheal tube is inserted and admitted to the cardiovascular surgery intensive care unit, and the endotracheal tube is removed in the intensive care unit.
* There is a clinical indication to perform lung expansion therapy
* Clear consciousness and able to cooperate with instructions

Exclusion Criteria:

* Hemodynamic instability (mean arterial pressure remains below 60 mmHg after infusion or vasopressor administration)
* Severe lung diseases (such as uncontrollable asthma, severe pulmonary obstruction, untreated pneumothorax, etc.)
* Unable to perform effective deep breathing (for example: vital capacity is less than 10 ml/kg or inspiratory capacity is less than 1/3 of the predicted value)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-06 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
The improvement of nursing staff's awareness rate of lung expansion therapy | week 2 after on-the-job training
  The improvement before and after on-the-job training
The improvement of nursing staff's correct rate of education of lung expansion therapy | week 2 after on-the-job training
  The improvement before and after on-the-job training

SECONDARY OUTCOMES:
The improvement of patients' correct rate of lung expansion therapy | week 2 after nurse staff's on-the-job training
  The improvement before and after nurse staff's on-the-job training
The improvement of respiratory complication rate | week 2 after nurse staff's on-the-job training
  The improvement before and after nurse staff's on-the-job training
Nurses' satisfaction of the quality improvement project survey | week 2 after nurse staff's on-the-job training
  Nurses' satisfaction of the quality improvement project

IPD SHARING:
Plan to Share IPD: No